CLINICAL TRIAL: NCT05826041
Title: Development, Implementation and Evaluation of an Integrated, Peer-Led, Group Intervention for Survivors of Domestic Violence
Brief Title: Project INSPIRE: INtervention Support Groups: Peers Inspiring Resilience and Empowerment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Site was unable to refer participants due to staffing issues post COVID
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000024110; 2018-SI-AX-0005 (Other Grant/Funding Number: Office on Violence Against Women (OVW))
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Domestic Violence
Keywords: Intimate Partner Violence

STUDY DESIGN:
Intervention Model Description: Other: INSPIRE support group Other: Intervention as usual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INSPIRE Group (Experimental): 90-minute support group; 9 content sessions over 18 weeks; co-led by a professional facilitator and peer.
  Interventions: Behavioral: (INSPIRE) INtervention Support groups: Peers Inspiring Resilience and Empowerment.
- Intervention as Usual: Traditional Domestic Violence Support Group (Active Comparator): 75-minute support group; 18-weeks; led by a domestic violence service provider counselor or advocate
  Interventions: Behavioral: Traditional Domestic Violence Support Group

INTERVENTIONS:
Behavioral: (INSPIRE) INtervention Support groups: Peers Inspiring Resilience and Empowerment. — The support group contains both structured components, which are psychoeducational and focused on skill-building, and an unstructured component where discussion is open and determined by the needs and interests of the clients present (e.g., support and process-oriented.)
  Arms: INSPIRE Group
Behavioral: Traditional Domestic Violence Support Group — The activities of the group are determined by agency staff from week to week and may be open group discussion, psychoeducation, or a combination of both.
  Arms: Intervention as Usual: Traditional Domestic Violence Support Group

SUMMARY:
The investigators will develop a new, integrated, group intervention to enhance safety, support, and empowerment for survivors of intimate partner violence in the community. The intervention will consist of 9 weekly, 90-minute group sessions that will teach specific skills for identifying various forms of trauma and abuse, developing mutually supportive relationships, safety planning and self-care, goal-oriented communication, empowerment and self-efficacy, goal setting, coping, and connecting to resources. The investigators will pilot test the intervention, including evaluating the process of implementation, including feasibility, acceptability/likeability, and safety, as well as evaluating outcomes of safety, support, and empowerment. Outcomes from the intervention will be compared to outcomes from a traditional domestic violence support group.

ELIGIBILITY:
Inclusion Criteria:

* Domestic Violence Service Provider client referred for support group services

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Intervention acceptability/likability: Participant ratings of group cohesion assessed using the Group Attitude Scale (GAS) | up to week 18
  Group cohesion will be assessed weekly by a modified version of the GAS. The 20 items are rated on a 1-5 Likert scale. A total score is computed by averaging the items. Scores range from 1-5, with higher scores indicating more group cohesion.
Intervention acceptability/likability: Participant ratings of acceptability assessed using the Trauma-Informed Practices Scale (TIPS) | 9 weeks
  Acceptability will be assessed using the Trauma-Informed Practices Scale (TIPS). TIPS is a 33-item self-report measure comprised of 6 subscales. This study will use 28 of the original 33 items representing 5 of the 6 subscales: agency, information, connection, strengths, and cultural responsiveness and inclusivity; the support for parenting subscale was excluded as the intervention is not designed specifically to support parents. Items are rated on a 0-3 Likert scale, and mean scores are computed for each subscale and overall scale. Scores range from 0-3, with higher scores representing perceived receipt of more trauma-informed services.
Intervention acceptability/likability: Participant ratings of acceptability assessed using the Trauma-Informed Practices Scale (TIPS) | 18 weeks
  Acceptability will be assessed using the Trauma-Informed Practices Scale (TIPS). TIPS is a 33-item self-report measure comprised of 6 subscales. This study will use 28 of the original 33 items representing 5 of the 6 subscales: agency, information, connection, strengths, and cultural responsiveness and inclusivity; the support for parenting subscale was excluded as the intervention is not designed specifically to support parents. Items are rated on a 0-3 Likert scale, and mean scores are computed for each subscale and overall scale. Scores range from 0-3, with higher scores representing perceived receipt of more trauma-informed services.
Intervention acceptability/likability: Participant ratings of Working alliance assessed using the Session Rating Scale (SRS) | up to week 18
  Working alliance will be measured using an adapted version of the SRS. The SRS is a 4-item visual analog instrument. Each item is assessed using a 0-10 point scale. This measure will be modified for the participant to rate the working alliance with the peer co-facilitator and professional co-facilitator separately, for a total of 6 questions. A total score is computed by summing each item. Scores will range from 0-60, with an overall score of less than 56, or 9 on any item, indicating potential concerns in working alliance
Change in safety-related empowerment assessed using the Measure of Victim Empowerment Related to Safety (MOVERS) Scale | Baseline, 9 weeks, 18 weeks
  Change in safety-related empowerment will be assessed using the Expectation of Support and Internal Tools subscales of the MOVERS Scale. Items are rated on a 1-5 Likert scale. Items corresponding to each subscale are averaged. Scores range from 1-5, with higher scores indicating higher levels of safety-related empowerment.
Change in support assessed using the Domestic Violence Resource Utilization (DVR) questionnaire | Baseline, 9 weeks, 18 weeks
  Change in support will be assessed using the DVR questionnaire. The 24 items represent various types of services/resources used, and a count variable (0-24) is computed to indicate the total number of different kinds of services/resources an individual use.
Change in social support assessed using the Medical Outcomes Study Social Support (MOS-SS) Survey | Baseline, 9 weeks, 18 weeks
  Change in support will be assessed using the MOS-SS Survey. The 19 items are rated on a 5-point Likert scale. Mean scores are computed for each of the four subscales (emotional/informational support, tangible support, affectionate support, and positive social interaction), and a total summary score. Scores range from 1-5, with higher scores indicating greater levels of support.
Change in empowerment assessed using the Personal Progress Scale - Revised (PPS-R) | Baseline, 9 weeks, 18 weeks
  Change in empowerment will be assessed using the PPS-R. The 28 items are rated on a 7-point Likert scale, and a total score is computed by averaging the items; total scores range from 1-7, with higher scores indicating higher levels of empowerment.

SECONDARY OUTCOMES:
Change in Wellbeing assessed using the Quality of Life questionnaire | Baseline, 9 weeks, 18 weeks
  Change in Wellbeing will be assessed using the Quality of Life questionnaire. The 9 items are rated on a 7-point Likert scale, and a total score is computed by averaging the items; total scores range from 1-7, with higher scores indicating higher levels of wellbeing.
Change in Wellbeing assessed using the Rosenberg Self-Esteem Scale | Baseline, 9 weeks, 18 weeks
  Change in Wellbeing will be assessed using the Rosenberg Self-Esteem Scale. The 10-item scale ranges from 0-30. Scores between 15 and 25 are within normal range; scores below 15 suggest low self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Tami P Sullivan, PhD, Principal Investigator — Department of Psychiatry, Yale School of Medicine
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No